CLINICAL TRIAL: NCT00189553
Title: A Multi-National,Randomized, Phase III, GCIG Intergroup Study Comparing Pegylated Liposomal Doxorubicin and Carboplatin Versus Paclitaxel and Carboplatin in Patients With Epithelial Ovarian Cancer in Late Relapse (> 6 Months)
Brief Title: Caelyx Plus Carboplatin Versus Paclitaxel Plus Carboplatin in Patients With Epithelial Ovarian Cancer in Late Relapse
Acronym: CALYPSO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Schering-Plough (Industry); Arbeitsgemeinschaft Gynaekologische Onkologie Austria (Other); AGO Study Group (Other); Australia New Zealand Gynaecological Oncology Group (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); NCIC Clinical Trials Group (Network); NSGO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALYPSO; EudraCT 2004-04456-39
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer
Keywords: Extra-ovarian papillary serous tumors; Relapse over 6 months; Previously received taxane derivative
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — liposomal doxorubicin; Carboplatin; Drugs, Generic; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (Active Comparator): Paclitaxel-Carboplatin
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Experimental (Experimental): Caelyx-Carboplatin
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Carboplatin

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — 30 mg/m² every 4 weeks during 6 cycles or until progression
  Other Names: Caelyx
  Arms: Experimental
Drug: Carboplatin — AUC 5 every 3/4 weeks during 6 cycles or until progression
  Other Names: generic drug
Drug: Paclitaxel — 175 mg/m² at day 1 every 3 weeks during 6 cycles or until progression
  Other Names: generic drug
  Arms: Standard

SUMMARY:
This is a study of the efficacy and safety of Caelyx (pegylated liposomal doxorubicin) in combination with carboplatin compared to the standard treatment of paclitaxel and carboplatin in patients with epithelial ovarian cancer in late relapse (> 6 months).

DETAILED DESCRIPTION:
The main purpose of this research study is to find out if treatment of late relapse of ovarian or fallopian tube or primary peritoneal cancer with liposomal doxorubicin (Caelyx) combined with carboplatin will control the tumor growth at least as well as standard treatment of paclitaxel and carboplatin. And it is hoped that substituting paclitaxel with Caelyx in combination with carboplatin will improve the tolerance of the treatment program with at least the same efficacy and fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18
* Histologically proven diagnosis of cancer of the ovary, the fallopian tube or extra-ovarian papillary serous tumors
* Measurable disease (Response Evaluation Criteria in Solid Tumor [RECIST] criteria) or cancer antigen (CA) 125 assessable disease (Gynecologic Cancer Intergroup [GCIG] criteria) or with histologically proven diagnosis of relapse
* Disease in progression > 6 months after a first or second platinum-based line. Patients should have previously received a taxane derivative.
* ECOG performance status < 2
* Life expectancy of at least 12 weeks
* Adequate bone marrow, renal, and hepatic function

Exclusion Criteria:

* Ovarian tumors of low malignant potential
* Non-epithelial ovarian or mixed epithelial/non-epithelial tumors
* Previous radiotherapy
* Prior diagnosis of malignancy
* Bowel obstruction, sub-occlusive disease, or presence of symptomatic brain metastases
* Pre-existing motor or sensory neurologic pathology or symptoms National Cancer Institute (NCI) - Common Terminology Criteria for Adverse Events (CTCAE) grade > 1
* History of congestive heart failure (New York Heart Association [NYHA] classification > 2), history of myocardial infarction within the last 6 months, or history of atrial or ventricular arrhythmias
* Severe active infection
* Severe hypersensitivity to products containing Cremophor EL and/or to compounds chemically related to paclitaxel, carboplatin or Caelyx
* Fertile women not using adequate contraceptive methods
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Actual)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of patients in both study groups | 5 years

SECONDARY OUTCOMES:
Qualitative and quantitative toxicities | 6 months
Quality of life | 6 months
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pujade-Lauraine, MD, PhD, Study Chair — GINECO GROUP
Locations (1):
- Hôpital Hôtel Dieu, Paris, France